CLINICAL TRIAL: NCT05850117
Title: Efficacies of Tetracycline-levofloxacin Quadruple Therapy, Standard Bismuth Quadruple Therapy and Amoxicillin-levofloxacin Quadruple Therapy in the Second-line Treatment of H Pylori Infection
Brief Title: Efficacies of Tetracycline-levofloxacin, Standard Bismuth, Amoxicillin-levofloxacin Quadruple Therapy for H.p
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, DENG-CHYANG WU, clinical professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20190136
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori Eradication
MeSH Terms: interventions — Esomeprazole; Tetracycline; Levofloxacin; Metronidazole; Amoxicillin

STUDY DESIGN:
Intervention Model Description: 1.Tetracycline combined with levofloxacin quadruple therapy 2. standard tincture quadruple therapy 2. amoxicillin combined with levofloxacin quadruple therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tetracycline combined with levofloxacin quadruple therapy (Active Comparator): esomeprazole 40mg twice a day + tripotassium dicitrate bismuthate 300mg four times a day+ tetracycline 500mg four times a day+ levofloxacin 500mg once a day
  Interventions: Drug: esomeprazole, tripotassium dicitrate bismuthate, tetracycline and levofloxacin
- standard tincture quadruple therapy (Active Comparator): esomeprazole 40mg twice a day + tripotassium dicitrate bismuthate 300mg four times a day
  + tetracycline 500mg four times a day + metronidazole 250mg four times a day
  Interventions: Drug: esomeprazole , tripotassium dicitrate bismuthate, tetracycline 500mg and metronidazole
- amoxicillin combined with levofloxacin quadruple therapy (Active Comparator): esomeprazole 40mg twice a day + tripotassium dicitrate bismuthate 300mg four times a day+ amoxicillin 500mg four times a day+ levofloxacin 500mg once a day
  Interventions: Drug: esomeprazole, tripotassium dicitrate bismuthate , amoxicillin and levofloxacin

INTERVENTIONS:
Drug: esomeprazole, tripotassium dicitrate bismuthate, tetracycline and levofloxacin — Tetracycline combined with levofloxacin quadruple therapy
  Arms: Tetracycline combined with levofloxacin quadruple therapy
Drug: esomeprazole , tripotassium dicitrate bismuthate, tetracycline 500mg and metronidazole — standard tincture quadruple therapy
  Arms: standard tincture quadruple therapy
Drug: esomeprazole, tripotassium dicitrate bismuthate , amoxicillin and levofloxacin — amoxicillin combined with levofloxacin quadruple therapy
  Arms: amoxicillin combined with levofloxacin quadruple therapy

SUMMARY:
1. Compare the efficacy of "Tetracycline combined with levofloxacin quadruple therapy", "standard tincture quadruple therapy" and "amoxicillin combined with levofloxacin quadruple therapy" on the second line of Helicobacter pylori sterilization.
2. To investigate the drug resistance of Helicobacter pylori and the host genotypes of CYP2C19 and IL-1B-511 on the sterilizing effect of three second-line Helicobacter pylori.

DETAILED DESCRIPTION:
The "standard tincture quadruple therapy" and the "proton pump inhibitor combined with fluoroquinolone and amoxicillin triple therapy" recommended by the 5th Mazdock-Florence Consensus Conference on the second line of Helicobacter pylori treatment The sterilization rate is not ideal (less than 80%). Recently, we have developed a "Tetracycline combined with levofloxacin quadruple therapy" for first-line treatment failure of H. pylori infection, with a relatively high sterilization rate (> 95%). A randomized controlled trial confirmed that the elimination rate of "Tetracycline combined with levofloxacin quadruple therapy" was better than "proton pump inhibitor combined with fluoroquinolone" after "standard triple therapy" and "non-tank tetratherapy" sterilization failure. Triple therapy with amoxicillin.

ELIGIBILITY:
Inclusion Criteria:

1. at least 20 years old
2. subject was failure for the first line therapy of Helicobacter pylori

Exclusion Criteria:

1. Those who are allergic to the drugs used in this study
2. Those who have had a stomach surgery
3. Those who have antibiotics within four weeks of treatment
4. Those who have severe cirrhosis, uremia or malignancy
5. Those who are a pregnant woman or a woman who breastfeeds

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the rate of Helicobacter pylori | 6 week after finish study drugs
  evalute eradication outcome by 13C urea breath test

SECONDARY OUTCOMES:
genotype analysis | 2 weeks after finishing study drgus
  CYP2C19 genotype, IL-1B-511 genotype

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan